CLINICAL TRIAL: NCT00528515
Title: Comparison of Desflurane and Propofol Anesthesia for Off-Pump Coronary Artery Bypass Grafting Surgery
Brief Title: Desflurane Versus Propofol Anesthesia for Off-Pump CABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Romuald Lango MD, PhD, Medical University of Gdańsk, Dept. of Cardiac Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AMG-NKEBN/364-A/2005
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Artery Disease
Keywords: anesthesia intravenous; propofol; anesthesia inhalation; desflurane; heart surgery; coronary artery by-pass off-pump; hemodynamic processes; anesthesia
MeSH Terms: conditions — Coronary Artery Disease | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): propofol
  Interventions: Drug: Diprivan (propofol), Astra-Zeneca
- 2 (Experimental): desflurane
  Interventions: Drug: Suprane (desflurane), Baxter

INTERVENTIONS:
Drug: Diprivan (propofol), Astra-Zeneca — continuous intravenous infusion with a dose of 3-5 mg/kg/h
  Other Names: propofol
  Arms: 1
Drug: Suprane (desflurane), Baxter — a vapor concentration of 3-7 vol% is maintained with use of vaporizer and under control of arterial blood pressure, heart rate, and BIS index.
  Other Names: desflurane
  Arms: 2

SUMMARY:
The purpose of this study is to prove if anesthesia maintained with the inhaled volatile anesthetic desflurane is superior to the intravenously applied propofol anesthesia in off-pump coronary artery bypass grafting (OP-CABG) surgery as measured by following parameters:

1. hemodynamic parameters during and after the operation,
2. pulmonary gas exchange, need for mechanical ventilation and for ICU and intrahospital stay,
3. release of heart muscle injury markers in response to surgery and intraoperative ischaemia,
4. inflammatory response to the operation.

We suspect that insufflation anesthesia with desflurane may be superior to intravenous anesthesia with propofol.

DETAILED DESCRIPTION:
General anesthesia will be induced by intravenous dosis of fentanyl, vecuronium and etomidate and further maintained either by inhaled desflurane or propofol infusion, with concomitant empirically administered fentanyl doses and continuous infusion of vecuronium.

After induction of anesthesia a Swan-Ganz catheter for continuous cardiac output, right ventricle end diastolic volume and blood saturation measurements will be introduced through the internal jugular vein. A transesophageal echocardiography probe will be placed additionally for the Tei-index measurement.

Hemodynamic parameters will be recorded at the following time points:

* before induction
* after induction
* during trachea intubation
* before skin incision
* 3 Min. after skin incision
* after sternotomy
* before heart positioning for graft placing
* before finishing placing each distal anastomoses
* 10, 20, 30, 40 min after placing the last anastomoses
* 10 Min. after admission to ICU, 6, 12, 18 and 24 hours after surgery.
* TEE measurements will be obtained after sternotomy and 20 Min after placing the last distal anastomoses.

The results will be compared while using the parametric ANOVA test for normally distributed continuous data or the nonparametric Kruskal-Wallis/Wilcoxon-U test for categoric or inhomogeneous distributed continuous data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease qualified for CABG off-pump surgery
* Elective surgery
* Signed informed consent

Exclusion Criteria:

* Left ventricle ejection fraction < 30%
* Serum creatinine > 2 mg/dL
* Emergency surgery
* Denied consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Markers of heart muscle injury and inflammation will be compared: troponin I, creatinine phosphokinase and its heart specific fraction, C-reactive protein. | within the first 2. days after surgery.

SECONDARY OUTCOMES:
Evidence of clinically definite heart infarct confirmed by ECG and/or echocardiography, and heart muscle specific creatinine phosphokinase increase. | To discharge from hospital (usually within 7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Lango, M.D., Ph.D., Study Director — Medical University of Gdańsk, Department of Cardiac Anesthesiology
Locations (1):
- Department of Cadiac Anesthesiology, Medical University of Gdańsk, Gdansk, Poland

REFERENCES:
- [Background] Xia Z, Luo T. Sevoflurane or desflurane anesthesia plus postoperative propofol sedation attenuates myocardial injury after coronary surgery in elderly high-risk patients. Anesthesiology. 2004 Apr;100(4):1038-9; author reply 1039-40. doi: 10.1097/00000542-200404000-00050. No abstract available. PMID 15087655
- [Background] Tritapepe L, Landoni G, Guarracino F, Pompei F, Crivellari M, Maselli D, De Luca M, Fochi O, D'Avolio S, Bignami E, Calabro MG, Zangrillo A. Cardiac protection by volatile anaesthetics: a multicentre randomized controlled study in patients undergoing coronary artery bypass grafting with cardiopulmonary bypass. Eur J Anaesthesiol. 2007 Apr;24(4):323-31. doi: 10.1017/S0265021506001931. Epub 2006 Dec 8. PMID 17156509
- [Background] Guarracino F, Landoni G, Tritapepe L, Pompei F, Leoni A, Aletti G, Scandroglio AM, Maselli D, De Luca M, Marchetti C, Crescenzi G, Zangrillo A. Myocardial damage prevented by volatile anesthetics: a multicenter randomized controlled study. J Cardiothorac Vasc Anesth. 2006 Aug;20(4):477-83. doi: 10.1053/j.jvca.2006.05.012. PMID 16884976
- [Background] De Hert SG, Cromheecke S, ten Broecke PW, Mertens E, De Blier IG, Stockman BA, Rodrigus IE, Van der Linden PJ. Effects of propofol, desflurane, and sevoflurane on recovery of myocardial function after coronary surgery in elderly high-risk patients. Anesthesiology. 2003 Aug;99(2):314-23. doi: 10.1097/00000542-200308000-00013. PMID 12883404
- [Derived] Mrozinski P, Lango R, Biedrzycka A, Kowalik MM, Pawlaczyk R, Rogowski J. Comparison of haemodynamics and myocardial injury markers under desflurane vs. propofol anaesthesia for off-pump coronary surgery. A prospective randomised trial. Anaesthesiol Intensive Ther. 2014 Jan-Mar;46(1):4-13. doi: 10.5603/AIT.2014.0002. PMID 24643920
- See also: Related Info — http://www.amg.gda.pl/uczelnia/informator/projekty.php?id=327